CLINICAL TRIAL: NCT05124405
Title: Monitoring Your Exercise-related Metrics Over Time Via Wearable Electronic Devices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0299; NCI-2019-02652 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2019-05-20; First posted 2021-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Diabetes
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart Rate Tracker (Fitbit) (Experimental): continuous heart rate activity
  Interventions: Other: Fitbit; Other: Continuous Glucose Monitor
- Continuous Glucose Monitor (CGM) (Experimental): monitoring daily exercise-related activities
  Interventions: Other: Fitbit; Other: Continuous Glucose Monitor

INTERVENTIONS:
Other: Fitbit — wearable activity tracker
Other: Continuous Glucose Monitor — wearable activity tracker

SUMMARY:
To test the use of a continuous activity and heart rate tracker (Fitbit) and continuous glucose monitor (CGM) in monitoring daily exercise-related activities.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the feasibility of a CGM-based physical activity intervention that includes the use of CGM and Fitbit®.

Secondary objectives:

To examine changes in physical activity motivation and other related psychosocial variables (e.g., intention, perceived benefits, outcome expectancy) before and after the intervention.

Exploratory objective:

Examine cancer-related biomarkers and their associations with daily glucose pattern.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old
* Body mass index (BMI) 25 kg/m2
* Engage in less than 150 minutes of moderate-intensity PA per week in the past month
* Capable of participating in moderate-vigorous unsupervised exercise (as determined by the Physical Activity Readiness Questionnaire (PARQ) or a medical release from their physician)
* Self-reported ability to walk one block without pain or discomfort
* Have a smart phone with daily internet access that is compatible with the LibreLink app
* Ability to speak, read, and write in English
* For the cancer survivor cohort (participant accession number #21 and beyond), individuals must have been diagnosed with stage I-III breast or colorectal cancer and completed adjuvant therapy (i.e., chemo and/or radiation therapy).

Exclusion Criteria:

* Self-reported current diagnosis or history of type 1 diabetes or type 2 diabetes
* Self-reported use of oral antidiabetic agents (OADs)
* Previous or current treatment with any insulin regimen other than basal insulin, e.g. prandial or pre-mixed insulin (short term treatment due to intercurrent illness including gestational is allowed at the discretion for the investigator)
* Current use of a continuous glucose monitor
* Fasting glucose > 125 mg/dL
* Pregnancy
* Self-reported health issues that limit physical activity
* On dialysis
* Work overnight shifts
* Unwilling to use CGM
* Current participation in other wellness or weight loss-related program or intervention
* Currently on a low-carb diet
* Unable to receive REDCap survey through their mobile phones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of the ( PA) Physical Activity intervention. | through study completion, an average of 1 year
  The use of CGM through the following criteria: CGM-specific refusal rate <20% at the participant recruitment phase and protocol adherence rates >80% at the end of the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Liao Y, Brannon GE, Rethorst CD, Baum M, Bevers TB, Schembre SM, Basen-Engquist KM. Using Continuous Glucose Monitoring as a Biological Feedback Strategy to Motivate Physical Activity in Cancer Survivors: A Mixed-Methods Pilot Study. Cancer Control. 2025 Jan-Dec;32:10732748251359406. doi: 10.1177/10732748251359406. Epub 2025 Jul 28. PMID 40719638
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org